CLINICAL TRIAL: NCT04315545
Title: Pregnancy Outcomes and Maternal Insulin Sensitivity
Acronym: PROMIS
Status: Terminated | Type: Observational
Why Stopped: slow recruitment, reached sufficient recruitment numbers for exploratory analysis
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, eline van der beek, Prof. dr. E.M. van der Beek, University Medical Center Groningen
Other Study IDs: 68845
Record Dates: First submitted 2020-02-20; First posted 2020-03-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes; Other "Heavy-For-Dates" Infants; Small for Gestational Age Infant; Diabetes Mellitus, Type 2
Keywords: Insulin sensitivity; Insulin insensitivity; Pregnancy; Metabolism; Neonatal outcomes; glucose metabolism; Oral glucose tolerance test; Meal tolerance test; neonatal health; maternal health; maternal insulin sensitivity; gestational weight gain; diagnostic tool; early screening; prevention; overweight; obesitiy; metabolic health; neonatal adiposity; maternal adiposity
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Insulin Resistance; Gestational Weight Gain; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples Without DNA — serum & plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy women pregnant of singleton with a BMI ≥25 kg/m2: Healthy women pregnant of singleton with a BMI ≥25 kg/m2 will be followed from 12 weeks of gestation till 6 months postpartum. Neonates will be followed from birth up to 6 months of age.
  Interventions: Diagnostic Test: meal tolerance test

INTERVENTIONS:
Diagnostic Test: meal tolerance test — In addition to the standard oral glucose tolerance (which is normally performed between 24-28 weeks of pregnancy), is used to test the metabolic resilience capacity of glucose, we will provide our participants with a different diagnostic tool named 'meal tolerance test' in an earlier stage of pregnancy (12-16 weeks), mid pregnancy (24-28 weeks) and 3 months postpartum.

SUMMARY:
The PROMIS study will focus on maternal insulin sensitivity thourghout pregnancy and postpartum in a moderate to high risk population (BMI ≥25 kg/m2) in developing adverse pregnancy outcomes. Next to the OGTT, the meal tolerance test (MTT) will be used as a tool for metabolic testing.

The investigators hypothesize that (early) pregnancy assessment of maternal glucose-insulin metabolism with a MTT in a moderate to high risk group identify more mothers at risk for adverse pregnancy outcomes compared with standard OGTT testing at 24-28 weeks.

DETAILED DESCRIPTION:
The worldwide prevalence of overweight and obesity is rapidly increasing, also affecting women of reproductive age. The prevalence of overweight women between 30-40 years in the Netherlands in 2017 was 39%. Women with a BMI ≥25 kg/m2 have excess adipose tissue which reduces insulin sensitivity and explains the correlated adverse outcomes for both mother and child.

Insulin sensitivity changes over the course of pregnancy due to the effect of placental hormones and is therefore normally decreased by the end of the second trimester to ensure a continuous supply of nutrients towards the growing fetus. Insulin resistance leads to beta-cell proliferation and larger volume of individual beta-cells, returning to non-pregnant levels after parturition. When beta-cell proliferation is not or inadequately increased, this may lead to hyperglycemia. It is shown that small increases in maternal glucose levels have a linear relationship with adverse outcomes. Maternal adverse outcomes are pre-eclampsia, caesarian section and gestational diabetes mellitus (GDM) on the short term and increased risk of weight retention and non-communicable diseases like cardiovascular diseases and diabetes mellitus type 2 (DM2) on the longer term. Adverse outcomes in infants are macrosomia, large for gestational age (LGA), small for gestational age (SGA) on the short term and a higher risk on childhood obesity and non-communicable diseases on the longer term. Adequate maternal insulin sensitivity throughout pregnancy is therefore critical.

Small maternal glucose increases could already be detected in an early stage of pregnancy. In the Netherlands hyperglycemia is standardly examined at the end of the second trimester in an at risk population by an oral glucose tolerance test (OGTT). This test is less suitable to detect mild hyperglycemia in early stages of pregnancy, with merely blood glucose levels as a result, and shows a lot of within subject variability. However markers of insulin sensitivity and related metabolic adaptations, for instance in lipid metabolism, may be a more straightforward measure that could potentially be detected earlier and allow for early intervention. An integration of postprandial responses of glucose/insulin following a meal challenge combined with lipid markers could provide clearer insights in maternal metabolic function. A test that could be used to examine this in more detail is a liquid meal tolerance test (MTT) which contains a balanced macro- and micronutrient composition. Assessing glucose homeostasis is not possible by only measuring glucose concentrations as there are numerous perturbations where glucose production and its utilization increases or decreases to the same extent without any changes in concentrations. For the understanding of the physiology and pathophysiology of glucose uptake and metabolism during pregnancy, glucose tracers should be followed.

The PROMIS study will specifically focus on the associations between insulin sensitivity in the mother in early pregnancy and fetal and neonatal outcomes with emphasis on growth and body composition. The investigators therefore hypothesize that when overweight pregnant women are challenged in early pregnancy with a MTT, the group of women with disturbed insulin sensitivity could be identified much earlier, and can therefore have a predictive role in adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton pregnant women (10-12 weeks of gestation)
* BMI ≥25 kg/m2
* FPG ≤7.0 mmol/l
* Dutch or English speaking
* Written informed consent

Exclusion Criteria:

* Serious health complications (Hypertension, Hyperlipidemia, Asthma, Haemochromatosis) or medication use that influence the glucose metabolism or fetal growth (e.g. corticosteroids).
* Multiple pregnancy
* pre-existing Diabetes type 1 and 2 defined as FPG ≥7.0 mmol/l or use of diabetes medication
* Participation in any other studies involving the investigation of medication or nutritional products or severe illness or antibiotic use in the two weeks prior to entry into the study
* HIV/Hepatitis
* Expectation of non-compliance to the study protocol, among others, a fear of needles
* Known allergies or intolerances for one or more nutritional ingredients in the MTT
* Psychological dysfunctions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population will be pregnant women with a BMI ≥25 kg/m2 with a moderate to high 'at risk' of developing gestational diabetes throughout pregnancy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
fasting glucose | T=0 min, before intake of test drink
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=10 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=20 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=30 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=45 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=60 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=90 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
postprandial glucose | T=120 min postprandial
  Bloood will be collected fasted and after intake of the MTT and OGTT
fasting and postprandial glucose | AUC and postprandial curve
  Bloood will be collected fasted and after intake of the MTT and OGTT
fasting insulin | T=0 min, before intake of test drink
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=10 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=20 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=30 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=45 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=60 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=90 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial insulin | T=120 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
fasting and postprandial insulin | AUC and postprandial curve
  Blood will be collected fasted and after intake of the MTT and OGTT

SECONDARY OUTCOMES:
Triglycerides | T=0 min, before intake of test drink
  Blood will be collected fasted
Total cholesterol | T=0 min, before intake of test drink
  Blood will be collected fasted
HDL-cholesterol | T=0 min, before intake of test drink
  Blood will be collected fasted
Free fatty acids | T=0 min, before intake of test drink
  Blood will be collected fasted
Hba1c | T=0 min, before intake of test drink
  Blood will be collected fasted
Fasting stable glucose isotopes | T=0, before intake of test drink
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=10 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=20 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=30 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=45 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=60 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=90 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
postprandial stable glucose isotopes | T=120 min postprandial
  Blood will be collected fasted and after intake of the MTT and OGTT
fasting and postprandial stable glucose isotopes | AUC and postprandial curve
  Blood will be collected fasted and after intake of the MTT and OGTT

OTHER OUTCOMES:
FFQ | between week 12-16 of gestation
  Food frequency questionnaire
FFQ | between 24-28 of gestation
  Food frequency questionnaire
FFQ | 1 month postpartum
  Food frequency questionnaire
FFQ | 3 months postpartum
  Food frequency questionnaire
AEBQ | between week 12-16 of gestation
  Adult eating behaviour questionnaire
AEBQ | between 24-28 of gestation
  Adult eating behaviour questionnaire
AEBQ | 1 month postpartum
  Adult eating behaviour questionnaire
AEBQ | 3 months postpartum
  Adult eating behaviour questionnaire
BEBQ | 1 month postpartum in child
  Baby eating behaviour questionnaire
BEBQ | 3 months postpartum in child
  Baby eating behaviour questionnaire
EQ | Between week 12-16 of gestation
  EQ-5D questionnaire
EQ | between week 24-28 of gestation
  EQ-5D questionnaire
EQ | 1 month postpartum
  EQ-5D questionnaire
EQ | 3 months postpartum
  EQ-5D questionnaire
PA | between week 12-16 of gestation
  Pregnancy physical activity questionnaire
PA | between week 24-28 of gestation
  Pregnancy physical activity questionnaire
PA | 1 month postpartum
  International physical activity questionnaire
PA | 3 months postpartum
  International physical activity questionnaire
MP | In week 24 of gestation
  Meal test preference questionnaire
MP | In week 25 of gestation
  Meal test preference questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eline M van der Beek, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Centre Groningen, Groningen
  - Medical Center Leeuwarden, Leeuwarden

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be submitted for publication in a peer reviewed journal
Supporting Information: Study Protocol
Time Frame: 2021 PROMIS design and study rationale published in Journal of Clinical Medicine
Access Criteria: access to detailed information by others will be subject to evaluation by the PI and project team, based on submission of an official request with details on what, why and how.

REFERENCES:
- [Background] Koning SH, Hoogenberg K, Lutgers HL, van den Berg PP, Wolffenbuttel BH. Gestational Diabetes Mellitus:current knowledge and unmet needs. J Diabetes. 2016 Nov;8(6):770-781. doi: 10.1111/1753-0407.12422. Epub 2016 Jul 28. PMID 27121958
- [Background] Venkataraman H, Ram U, Craik S, Arungunasekaran A, Seshadri S, Saravanan P. Increased fetal adiposity prior to diagnosis of gestational diabetes in South Asians: more evidence for the 'thin-fat' baby. Diabetologia. 2017 Mar;60(3):399-405. doi: 10.1007/s00125-016-4166-2. Epub 2016 Dec 2. PMID 27913848
- [Background] World Health Organization. World health statistics 2016: Monitoring health for the SDGs sustainable development goals. World Health Organization; 2016.
- [Background] Ko GT, Chan JC, Woo J, Lau E, Yeung VT, Chow CC, Cockram CS. The reproducibility and usefulness of the oral glucose tolerance test in screening for diabetes and other cardiovascular risk factors. Ann Clin Biochem. 1998 Jan;35 ( Pt 1):62-7. doi: 10.1177/000456329803500107. PMID 9463740
- [Background] Maegawa Y, Sugiyama T, Kusaka H, Mitao M, Toyoda N. Screening tests for gestational diabetes in Japan in the 1st and 2nd trimester of pregnancy. Diabetes Res Clin Pract. 2003 Oct;62(1):47-53. doi: 10.1016/s0168-8227(03)00146-3. PMID 14581157
- [Background] Seshiah V, Cynthia A, Balaji V, Balaji MS, Ashalata S, Sheela R, Thamizharasi M, Arthi T. Detection and care of women with gestational diabetes mellitus from early weeks of pregnancy results in birth weight of newborn babies appropriate for gestational age. Diabetes Res Clin Pract. 2008 May;80(2):199-202. doi: 10.1016/j.diabres.2007.12.008. Epub 2008 Feb 4. PMID 18249458
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Chen C, Xu X, Yan Y. Estimated global overweight and obesity burden in pregnant women based on panel data model. PLoS One. 2018 Aug 9;13(8):e0202183. doi: 10.1371/journal.pone.0202183. eCollection 2018. PMID 30092099
- [Background] Catalano PM, Ehrenberg HM. The short- and long-term implications of maternal obesity on the mother and her offspring. BJOG. 2006 Oct;113(10):1126-33. doi: 10.1111/j.1471-0528.2006.00989.x. Epub 2006 Jul 7. PMID 16827826
- [Background] Zhu Y, Zhang C. Prevalence of Gestational Diabetes and Risk of Progression to Type 2 Diabetes: a Global Perspective. Curr Diab Rep. 2016 Jan;16(1):7. doi: 10.1007/s11892-015-0699-x. PMID 26742932
- [Background] Koning SH, van Zanden JJ, Hoogenberg K, Lutgers HL, Klomp AW, Korteweg FJ, van Loon AJ, Wolffenbuttel BHR, van den Berg PP. New diagnostic criteria for gestational diabetes mellitus and their impact on the number of diagnoses and pregnancy outcomes. Diabetologia. 2018 Apr;61(4):800-809. doi: 10.1007/s00125-017-4506-x. Epub 2017 Nov 22. PMID 29167927
- [Background] Koning SH, Hoogenberg K, Scheuneman KA, Baas MG, Korteweg FJ, Sollie KM, Schering BJ, van Loon AJ, Wolffenbuttel BH, van den Berg PP, Lutgers HL. Neonatal and obstetric outcomes in diet- and insulin-treated women with gestational diabetes mellitus: a retrospective study. BMC Endocr Disord. 2016 Sep 29;16(1):52. doi: 10.1186/s12902-016-0136-4. PMID 27680327
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Feig DS, Zinman B, Wang X, Hux JE. Risk of development of diabetes mellitus after diagnosis of gestational diabetes. CMAJ. 2008 Jul 29;179(3):229-34. doi: 10.1503/cmaj.080012. PMID 18663202
- [Background] Yang X, Hsu-Hage B, Zhang H, Zhang C, Zhang Y, Zhang C. Women with impaired glucose tolerance during pregnancy have significantly poor pregnancy outcomes. Diabetes Care. 2002 Sep;25(9):1619-24. doi: 10.2337/diacare.25.9.1619. PMID 12196437
- [Background] Langer O, Umans JG, Miodovnik M. The proposed GDM diagnostic criteria: a difference, to be a difference, must make a difference. J Matern Fetal Neonatal Med. 2013 Jan;26(2):111-5. doi: 10.3109/14767058.2012.734874. Epub 2012 Oct 30. PMID 23039192
- [Background] Hadlock FP, Harrist RB, Sharman RS, Deter RL, Park SK. Estimation of fetal weight with the use of head, body, and femur measurements--a prospective study. Am J Obstet Gynecol. 1985 Feb 1;151(3):333-7. doi: 10.1016/0002-9378(85)90298-4. PMID 3881966
- [Background] Ferrara A, Peng T, Kim C. Trends in postpartum diabetes screening and subsequent diabetes and impaired fasting glucose among women with histories of gestational diabetes mellitus: A report from the Translating Research Into Action for Diabetes (TRIAD) Study. Diabetes Care. 2009 Feb;32(2):269-74. doi: 10.2337/dc08-1184. Epub 2008 Nov 4. PMID 18984776
- [Background] Malcolm J, Lawson ML, Gaboury I, Keely E. Risk perception and unrecognized type 2 diabetes in women with previous gestational diabetes mellitus. Obstet Med. 2009 Sep;2(3):107-10. doi: 10.1258/om.2009.080063. Epub 2009 Sep 1. PMID 27582823
- [Background] Noctor E, Dunne FP. Type 2 diabetes after gestational diabetes: The influence of changing diagnostic criteria. World J Diabetes. 2015 Mar 15;6(2):234-44. doi: 10.4239/wjd.v6.i2.234. PMID 25789105
- [Background] Cobelli C, Man CD, Sparacino G, Magni L, De Nicolao G, Kovatchev BP. Diabetes: Models, Signals, and Control. IEEE Rev Biomed Eng. 2009 Jan 1;2:54-96. doi: 10.1109/RBME.2009.2036073. PMID 20936056
- [Background] Sonagra AD, Biradar SM, K D, Murthy D S J. Normal pregnancy- a state of insulin resistance. J Clin Diagn Res. 2014 Nov;8(11):CC01-3. doi: 10.7860/JCDR/2014/10068.5081. Epub 2014 Nov 20. PMID 25584208
- [Background] Catalano PM, Huston L, Amini SB, Kalhan SC. Longitudinal changes in glucose metabolism during pregnancy in obese women with normal glucose tolerance and gestational diabetes mellitus. Am J Obstet Gynecol. 1999 Apr;180(4):903-16. doi: 10.1016/s0002-9378(99)70662-9. PMID 10203659
- [Background] Lain KY, Catalano PM. Metabolic changes in pregnancy. Clin Obstet Gynecol. 2007 Dec;50(4):938-48. doi: 10.1097/GRF.0b013e31815a5494. PMID 17982337
- [Background] Catalano PM, Kirwan JP, Haugel-de Mouzon S, King J. Gestational diabetes and insulin resistance: role in short- and long-term implications for mother and fetus. J Nutr. 2003 May;133(5 Suppl 2):1674S-1683S. doi: 10.1093/jn/133.5.1674S. PMID 12730484